CLINICAL TRIAL: NCT01468766
Title: Effects of a Supervised Progressive Resistance Training With Breast Cancer Patients During Adjuvant Radiotherapy - A Randomised Controlled Intervention Trial
Brief Title: Effects of a Supervised Progressive Resistance Training With Breast Cancer Patients During Adjuvant Radiotherapy
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other); National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Principal Investigator, Karen Steindorf, Prof. Dr. Karen Steindorf / Dr. Karin Potthoff, National Center for Tumor Diseases, Heidelberg, German Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEST
Record Dates: First submitted 2011-10-11; First posted 2011-11-09 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer; Cancer-related Fatigue
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Resistance training (Active Comparator)
  Interventions: Other: Supervised progressive resistance training
- Relaxation training (Active Comparator)
  Interventions: Other: Supervised progressive muscle relaxation training (Jacobson method)

INTERVENTIONS:
Other: Supervised progressive resistance training — 2x60 minutes per week for 12 weeks
  Arms: Resistance training
Other: Supervised progressive muscle relaxation training (Jacobson method) — 2x60 minutes per week for 12 weeks
  Arms: Relaxation training

SUMMARY:
The purpose of this randomized intervention study is to investigate the effects and biological mechanisms of a supervised 12-week progressive resistance training on fatigue and immunological and inflammatory biomarkers in breast cancer patients during adjuvant radiotherapy. To determine the effect of the exercise itself beyond potential psychosocial effects due to attention by trainers or the group support, patients in the control group have a comparable training schedule (i.e. 60 min, twice a week, for 12 weeks) but with relaxation training (Jacobsen method).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed primary breast cancer, stage I-III, after lumpectomy or mastectomy, indication for adjuvant radiotherapy
* BMI: 18-40
* ability to understand and follow the study protocol

Exclusion Criteria:

* contraindication for exercise
* participation in the BEATE trial or another systematic resistance or relaxation training

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Fatigue measured by Fatigue Assessment Questionnaire (FAQ) | change between baseline and week 13 (end of intervention)

SECONDARY OUTCOMES:
Quantity of FoxP3+ CD25+ regulatory T-cells | change between baseline and week 13 (end of intervention)
Inflammatory parameter CRP, SAA and IL-6 | change between baseline and week 13 (end of intervention)
Circulating lymphocytes subpopulations (CD4+, CD8+, CD56+) | change between baseline and week 13 (end of intervention)
Specificity of FoxP3+ CD25+ regulatory T-cells (in a subgroup only) | change between baseline and week 13 (end of intervention)
  immunmagnetic purification of the Treg (Selection by CD4 und CD25 expression; MACS-beads) by co-culturing of titrated Treg with 3H marked autologuous, polyclonal (anti CD3/CD28) activiated, conventional T-cells (CD4+, CD25+) and subsequent assessment of the proliferation of conventional T-cells.
  Zur Bestimmung der Treg-Spezifität wurde eigens eine neue Methode entwickelt, die auf der signifikant erhöhten suppressiven Aktivität antigenspezifisch aktivierter Treg, gegenüber nicht aktivierten Treg, basiert.
Quality of Life measured by the European Organisation for Research and Treatment of Cancer questionnaire (EORTC-QLQ30/BR23) | change between baseline and week 13 (end of intervention)
Depression measured by "Allgemeine Depressionsskala" (ADS, the German version of the Center for Epidemiological Studies Depression Scale (CES-D)) | change between baseline and week 13 (end of intervention)
Muscle strength measured at the IsoMed2000® | change between baseline and week 13 (end of intervention)
Cardiorespiratory fitness measured by ergospirometry | change between baseline and week 13 (end of intervention)
Number of participants with lymphedema, pain, nausea, dyspnea, or tachycardia as a measure of safety of resistance training during radiotherapy. | events with onset or worsening during the 12-week intervention period are considered
Cognitive performance measured by the Trail-Making-Test | change between baseline and week 13 (end of intervention)
Toxicity of radiotherapy (acute radio dermatitis; LENT-SOMA classification for late effects) | acute toxicity during radio therapy and late effects 6 weeks after end of radio therapy are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center; Karin Potthoff, Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- National Center for Tumor Diseases, Heidelberg, Germany

REFERENCES:
- [Background] Potthoff K, Schmidt ME, Wiskemann J, Hof H, Klassen O, Habermann N, Beckhove P, Debus J, Ulrich CM, Steindorf K. Randomized controlled trial to evaluate the effects of progressive resistance training compared to progressive muscle relaxation in breast cancer patients undergoing adjuvant radiotherapy: the BEST study. BMC Cancer. 2013 Mar 28;13:162. doi: 10.1186/1471-2407-13-162. PMID 23537231
- [Result] Steindorf K, Schmidt ME, Klassen O, Ulrich CM, Oelmann J, Habermann N, Beckhove P, Owen R, Debus J, Wiskemann J, Potthoff K. Randomized, controlled trial of resistance training in breast cancer patients receiving adjuvant radiotherapy: results on cancer-related fatigue and quality of life. Ann Oncol. 2014 Nov;25(11):2237-2243. doi: 10.1093/annonc/mdu374. Epub 2014 Aug 5. PMID 25096607
- [Result] Klassen O, Schmidt ME, Scharhag-Rosenberger F, Sorkin M, Ulrich CM, Schneeweiss A, Potthoff K, Steindorf K, Wiskemann J. Cardiorespiratory fitness in breast cancer patients undergoing adjuvant therapy. Acta Oncol. 2014 Oct;53(10):1356-65. doi: 10.3109/0284186X.2014.899435. Epub 2014 May 16. PMID 24837860
- [Result] Schmidt ME, Meynkohn A, Habermann N, Wiskemann J, Oelmann J, Hof H, Wessels S, Klassen O, Debus J, Potthoff K, Steindorf K, Ulrich CM. Resistance Exercise and Inflammation in Breast Cancer Patients Undergoing Adjuvant Radiation Therapy: Mediation Analysis From a Randomized, Controlled Intervention Trial. Int J Radiat Oncol Biol Phys. 2016 Feb 1;94(2):329-37. doi: 10.1016/j.ijrobp.2015.10.058. Epub 2015 Nov 2. PMID 26853341
- [Result] Gollhofer SM, Wiskemann J, Schmidt ME, Klassen O, Ulrich CM, Oelmann J, Hof H, Potthoff K, Steindorf K. Factors influencing participation in a randomized controlled resistance exercise intervention study in breast cancer patients during radiotherapy. BMC Cancer. 2015 Mar 27;15:186. doi: 10.1186/s12885-015-1213-1. PMID 25885634
- [Result] Scharhag-Rosenberger F, Kuehl R, Klassen O, Schommer K, Schmidt ME, Ulrich CM, Wiskemann J, Steindorf K. Exercise training intensity prescription in breast cancer survivors: validity of current practice and specific recommendations. J Cancer Surviv. 2015 Dec;9(4):612-9. doi: 10.1007/s11764-015-0437-z. Epub 2015 Feb 26. PMID 25711667
- [Result] Schmidt ME, Semik J, Habermann N, Wiskemann J, Ulrich CM, Steindorf K. Cancer-related fatigue shows a stable association with diurnal cortisol dysregulation in breast cancer patients. Brain Behav Immun. 2016 Feb;52:98-105. doi: 10.1016/j.bbi.2015.10.005. Epub 2015 Oct 9. PMID 26456694
- [Derived] Koeppel M, Steindorf K, Schmidt ME, Rosenberger F, Wiskemann J. Variability in resistance training trajectories of breast cancer patients undergoing therapy. Support Care Cancer. 2024 Dec 10;33(1):12. doi: 10.1007/s00520-024-09001-4. PMID 39656317
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Schmidt ME, Chong M, Klassen O, Wiskemann J, Steindorf K. Longitudinal associations of bioelectrical phase angle and fatigue in breast cancer patients. Int J Cancer. 2023 Sep 15;153(6):1192-1200. doi: 10.1002/ijc.34630. Epub 2023 Jun 20. PMID 37337948
- [Derived] Steindorf K, Wiskemann J, Ulrich CM, Schmidt ME. Effects of exercise on sleep problems in breast cancer patients receiving radiotherapy: a randomized clinical trial. Breast Cancer Res Treat. 2017 Apr;162(3):489-499. doi: 10.1007/s10549-017-4141-8. Epub 2017 Feb 8. PMID 28181128